CLINICAL TRIAL: NCT02265666
Title: Randomised, Open-label, Two-way Crossover Study in Male Healthy Volunteers to Investigate the Relative Bioavailability of BIIL 284 BS 5 mg Tablet FF in Comparison to Tablet C After Ingestion of a Standardised Meal
Brief Title: Relative Bioavailability, Safety and Tolerability of Two Tablet Formulations of BIIL 284 BS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 543.31
Record Dates: First submitted 2014-10-15; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- BIIL 284 BS Tablet FF (Experimental)
  Interventions: Drug: BIIL 284 BS Tablet FF; Other: standard breakfast
- BIIL 284 BS tablet C (Active Comparator)
  Interventions: Drug: BIIL 284 BS tablet C; Other: standard breakfast

INTERVENTIONS:
Drug: BIIL 284 BS Tablet FF
  Arms: BIIL 284 BS Tablet FF
Drug: BIIL 284 BS tablet C
  Arms: BIIL 284 BS tablet C
Other: standard breakfast

SUMMARY:
The objective of the present study is to investigate the relative bioavailability of BIIL 284 BS Tablet FF in comparison to the tablet C at a dose of 5 mg after a standard breakfast in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* All participants are healthy males
* Age range from 21 to 50 years
* Broca-Index: within +- 20% of normal weight
* In accordance with Good Clinical Practice (GCP) and local legislation each volunteer is supposed to give their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrollment in the study
* Use of any drugs which might influence the results of the trial (<= one week prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60g/day)
* Drug abuse
* Blood donation (>= 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within the last week before the study )
* Any laboratory value outside the reference range of clinical relevance

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2001-10; Primary Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours after drug administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 24 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 24 hours after drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 24 hours after drug administration
Terminal rate constant in plasma | up to 24 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 24 hours after drug administration
MRTtot (total mean residence time) | up to 24 hours after drug administration
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) | up to 24 hours after drug administration
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | up to 24 hours after drug administration
Number of subjects with adverse events | up to 8 days after last drug administration
Number of subjects with clinically significant findings in vital functions | up to 8 days after last drug administration
  blood pressure, pulse rate, ECG
Number of subjects with clinically significant findings in laboratory tests | up to 8 days after last drug administration